CLINICAL TRIAL: NCT04863261
Title: Facilitating the Management of CAB+RPV LA Patient Visits Through Daily Alerts and Morning Huddles
Brief Title: Cabenuva Injection Tracking in CHORUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epividian (Industry)
Collaborators: AIDS Healthcare Foundation (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00050130
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial. The clinics will be randomized to either start using the Cabenuva Scheduling Alerts in the Retention & Huddle modules of the CHORUS App (Intervention Arm) or to standard of care (Control Arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Clinics randomized to the intervention. A notification will be sent to the provider when a patient on CAB+RPV LA needs to be scheduled for their injections or when an appointment needs to be confirmed. Alerts are sent out to the provider when a patient is due or overdue for their injections.
  Interventions: Other: Cabenuva Scheduling Alerts in the Retention & Huddle modules of the CHORUS App
- Control (No Intervention): Clinics randomized to the control group. No alerts or notification will be sent. The providers will manage their CAB+RPV LA patients using standard of care in their clinic.

INTERVENTIONS:
Other: Cabenuva Scheduling Alerts in the Retention & Huddle modules of the CHORUS App — The CHORUS App has been developed as a tool for clinicians to easily visualize important patient information from their smart phones. Relevant information is electronically distributed and placed within the corresponding module in the CHORUS HCP mobile app for iOS and Android.
  Arms: Intervention

SUMMARY:
This is a cluster randomized trial in which clinics will be randomized to the intervention or the control arm. The purpose of this study is to assess if receiving alerts can help providers manage the scheduling of monthly cabotegravir + rilpivirine long-acting injections for the treatment of HIV.

DETAILED DESCRIPTION:
A novel long-acting HIV antiretroviral therapy has recently been approved by the FDA: cabotegravir and rilpivirine delivered through intramuscular injection. These injections should be administered monthly, on the same day of the month as the initiation injections, up to 7 days before or after the date of the scheduled monthly injection visit.

This is a cluster randomized trial in which clinics will be randomized to the intervention or the control arm. Providers in the intervention group will receive alerts to remind them when patients are due for their injections, or if they missed their treatment window. Providers in the control group will not receive alerts and will manage injections as per their clinic's standard process. Surveys will be administered to understand the utility of the alerts for the management of these injections.

ELIGIBILITY:
Inclusion Criteria (patients):

* As per label, routine clinical care

Inclusion Criteria (clinics):

* AIDS Healthcare Foundation (AHF) Clinic
* HIV primary care clinic
* Minimum of 100 people living with HIV in care with a viral load <50 copies/mL at the time of randomization (satellites will be included in the count of their parent clinic).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment-window | 9 months
  Patient returns for their injections +/- 7 days from target date
Acceptability and usefulness of the intervention | Month 1
  Survey to assess the implementation of the Cabenuva Scheduling Alerts in the Retention & Huddle modules of the CHORUS App.
Acceptability and usefulness of the intervention | Month 9
  Survey to assess the implementation of the Cabenuva Scheduling Alerts in the Retention & Huddle modules of the CHORUS App.

SECONDARY OUTCOMES:
Number of CAB+RPV LA patients managed through the app | 9 months
  Reach
Number of clinics that use the App for the management of CAB+RPV LA patients | 9 month
  Adoption

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wohlfeiler, MD, Principal Investigator — AHF
Locations (1):
- AIDS Healthcare Foundation, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wohlfeiler MB, Brunet L, Cochran Q, Fusco JS, Hsu RK, Fusco GP. Improving Adherence to the Target Window for Cabotegravir + Rilpivirine Long-Acting Injections Through the CHORUS App and Web Portal: A Cluster Randomized Trial. J Int Assoc Provid AIDS Care. 2024 Jan-Dec;23:23259582241245223. doi: 10.1177/23259582241245223. PMID 38613372